CLINICAL TRIAL: NCT06204575
Title: Focused Ultrasound Thalamotomy for Tremor Relief in Atypical Parkinsonism
Acronym: FUSAP
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ilana Schlesinger, Director Movement Disorders Institute, clinical senior lecturer, Chair of Neurology, Rappaport Faculty of Medicine, Technion-Israel Institute of Technology Haifa, Israel, Rambam Health Care Campus
Other Study IDs: RMB-0404-17
Record Dates: First submitted 2023-12-31; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Atypical Parkinsonism; Dementia With Lewy Bodies; Multiple System Atrophy, MSA
Keywords: focused ultrasound; tremor; surgery; thalamotomy
MeSH Terms: conditions — Lewy Body Disease; Multiple System Atrophy; Thyroid Dyshormonogenesis 2A; Tremor | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
The goal of this retrospective observational study is to describe the efficacy of focused ultrasound ventral-intermediate nucleus thalamotomy in patients with atypical parkinsonism.

* Is this treatment efficacious in patients with multiple system atrophy?
* Is this treatment efficacious in patients with diffuse Lewy Body Dementia? Data will be collected from patients charts.

ELIGIBILITY:
Inclusion Patients that underwent FUS ventral-intermediate nucleus thalamotomy Suffer from multiple system atrophy-Parkinsonian type (MSA-P) or dementia with Lewy bodies (DLBD).

-

Exclusion Criteria:

* Patients that did not underwent FUS ventral-intermediate nucleus thalamotomy
* Patients that underwent FUS ventral-intermediate nucleus thalamotomy and do not suffer from MSA or DLBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent FUS VIM-thalamotomy and suffered from MSA or DLBD
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor | baseline, pre-procedure, 1 month, 6 months and 1 year following procedure
  tremor assessment by Clinical Rating Scale for Tremor. Scores ranging from 0 to 156, with higher scores indicating more severe tremor.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided